CLINICAL TRIAL: NCT04110054
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-selection Study of S-600918 in Patients With Refractory Chronic Cough
Brief Title: Evaluation of S-600918 in Adults With Refractory Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1812VA323
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Chronic Cough
Keywords: P2X3 receptor antagonist; Refractory chronic cough; S-600918
MeSH Terms: conditions — Chronic Cough | interventions — sivopixant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- S-600918 50 mg (Experimental): Participants will receive 50 mg S-600918 orally once a day for 28 days.
  Interventions: Drug: S-600918
- S-600918 150 mg (Experimental): Participants will receive 150 mg S-600918 orally once a day for 28 days.
  Interventions: Drug: S-600918
- S-600918 300 mg (Experimental): Participants will receive 300 mg S-600918 orally once a day for 28 days.
  Interventions: Drug: S-600918
- Placebo (Placebo Comparator): Participants will receive placebo to S-600918 orally once a day for 28 days.
  Interventions: Drug: Placebo to S-600918

INTERVENTIONS:
Drug: S-600918 — Tablets for oral administration
  Other Names: Sivopixant
  Arms: S-600918 150 mg; S-600918 300 mg; S-600918 50 mg
Drug: Placebo to S-600918 — Tablets for oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the optimal dose of S-600918 in patients with refractory chronic cough by evaluating the change from baseline in 24-hour cough frequency (coughs per hour) with S-600918 compared with placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Having refractory chronic cough (including unexplained chronic cough) for at least 1 year.
* If female and of childbearing potential, agreement to use one of the allowed contraceptive methods.
* Capable of giving signed informed consent.

Key Exclusion Criteria:

* Currently smokes or uses potentially irritating inhalational agents (eg, e-cigarettes, smokeless cigarettes, vaping); stopped smoking or using potentially irritating inhalational agents within the last year; or has a smoking history of 20 pack-years or more.
* Has chronic obstructive pulmonary disease or uncontrolled asthma.
* Has a clinically unstable medical condition.
* History of or ongoing significant psychiatric disorder.
* History of respiratory tract infection or significant change in lung function or a pulmonary condition in the last 4 weeks.
* History of malignancy in the last 5 years.
* History of severe drug allergy.
* History of alcohol or drug abuse in the last year or currently uses any form of marijuana or illicit drugs.
* Has a clinically significant finding on a chest x-ray or chest computed tomography (CT) scan in the last year.
* Has systolic blood pressure > 160 mm Hg or diastolic blood pressure > 90 mm Hg.
* Received S-600918 previously.
* Received an investigational drug in the last 3 months.
* Received an angiotensin converting enzyme (ACE) inhibitor in the last 3 months or requires such treatment.
* Has a positive serologic test for human immunodeficiency virus (HIV) antigen or antibody, hepatitis B virus surface antigen, or hepatitis C virus ribonucleic acid (RNA).
* If female, pregnant or trying to become pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (136):
- United States (51):
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Alliance for Multispecialty Research, Tempe, Arizona
  - Southern California Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Allergy & Asthma Associates of Southern California dba Southern California Research, Mission Viejo, California
  - California Medical Research Associates, Inc., Northridge, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Institute of HealthCare Assessment, Inc., San Diego, California
  - Sher Allergy Specialist/Center for Cough, Largo, Florida
  - Medical Research Of Central Florida, LLC, Leesburg, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - University of Kansas Medical Center-Hospital, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Abraham Research PLLC, Fort Mitchell, Kentucky
  - Shionogi Research Site, Bangor, Maine
  - St. Joseph's Hospital, Bangor, Maine
  - Minnesota Lung Center, Edina, Minnesota
  - Mayo Clinic Pulmonary Clinical Research Unit, Rochester, Minnesota
  - Mayo Clinic, Division of Pulmonary and Critical Care Medicine, Rochester, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - University of Missouri Hospital and Clinics, ENT & Allergy Center of Missouri, Columbia, Missouri
  - University of Missouri Hospital and Clinics, Hearing and Balance Center, Columbia, Missouri
  - University of Missouri Hospital - Clinical Research Center, Columbia, Missouri
  - Clayton Sleep Institute, LLC, St Louis, Missouri
  - Associated Specialists in Medicine, PC, St Louis, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Creighton University Clinical Research Office, Omaha, Nebraska
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - American Health Research Inc, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Northwest Research Center, Portland, Oregon
  - Clinical Research Associates of Central PA, LLC, DuBois, Pennsylvania
  - AAPRI Clinical Research Institute, Warwick, Rhode Island
  - ADAC Research, PA, Greenville, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Pharmaceutical Research & Consulting, Inc, Dallas, Texas
  - MCA Research, Houston, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Allergy and Asthma Care of Waco, Waco, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Intermountain Clinical Research, Draper, Utah
  - Tidewater Physicians Multispecialty Group Clinical Research, Williamsburg, Virginia
  - Allergy, Asthma & Sinus Center, S.C., Greenfield, Wisconsin
- Czechia (6):
  - Fakultní Nemocnice Olomouc, Olomouc, Czech Republic
  - MUDr. I. Čierná-Peterová s.r.o., Brandýs nad Labem-Stará Boleslav
  - Plicní Ambulance Rokycany s.r.o., Rokycany
  - MUDr. Jaroslav Mareš -, Strakonice
  - Plicní středisko Teplice s.r.o., Teplice
  - Pneumologie Varnsdorf s.r.o., Varnsdorf
- Japan (38):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukui Prefectural Hospital, Fukui-shi, Fukui
  - Kyushu Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuoka, Fukuoka
  - Nishi Fukuoka Hospital, Fukuoka, Fukuoka
  - Iizuka Hospital, Iizuka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Tohno Chuo Clinic, Mizunami-shi, Gifu
  - Mazda Hospital of Mazda Motor Corporation, Aki-gun, Hiroshima
  - Japan Mutual Aid Association of Public School Teachers Chugoku Central Hospital, Fukuyama, Hiroshima
  - Makita Hospital, Sapporo, Hokkaido
  - Idaimae Minamiyojo Int Clinic, Sapporo, Hokkaido
  - Nakatani Hospital, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Hitachi, Ltd. Hitachinaka General Hospital, Hitachi-Naka, Ibaraki
  - National Hospital Organization Ibarakihigashi National Hospital, Naka-gun, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Sakaide City Hospital, Sakaide-shi, Kagawa-ken
  - Kamei Internal Medicine and Respiratory Clinic, Takamatsu, Kagawa-ken
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - National Hospital Organization Sagamihara National Hospital, Sagamihara-shi, Kanagawa
  - Kaiseikai Kita Shin Yokohama Internal Medicine Clinic, Yokohama, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tohoku Rosai Hospital, Sendai, Miyagi
  - Lee's Clinic, Osaka, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai-shi, Osaka
  - Japan Organization of Occupational Health and Safety Hamamatsu Rosai Hospital, Hamamatsu, Shizuoka
  - Shizuoka General Hospital, Shizuoka, Shizuoka
  - Nihonbashi Medical & Allergy Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Takahashi Medical Clinic, Kokubunji-shi, Tokyo
  - Senzoku Kokyuuki Allergy Clinic, Ōta-ku, Tokyo
  - Yoga Allergy Clinic, Setagaya City, Tokyo
  - KONO Medical Clinic, Setagaya-ku, Tokyo
  - Koukokukai Ebisu Clinic, Shibuya-shi, Tokyo
  - Tokyo Shinagawa Hospital Medical Corporation Association Tokyokyojuno-kai, Shinagawa-ku, Tokyo
  - Kouwakai Kouwa Clinic, Toshima-ku, Tokyo
  - Shimonoseki City Hospital, Shimonoseki-shi, Yamaguchi
- Poland (13):
  - Prywatny Gabinet lnternistyczno-Alergologiczny, Bialystok
  - Centrum Medycyny Oddechowej Mroz sp. j., Bialystok
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Centrum Medyczne Silmedic Sp. z o. o., Katowice
  - Gyncentrum Sp. Z o. o., Katowice
  - Diamond Clinic, Krakow
  - Poradnia Alergologiczna SPZOZ USK nr 1 UM w Lodzi, Lodz
  - Ostrowieckie CM S.C. A. Olech-Cudzik, K. Cudzik, Ostrowiec Świętokrzyski
  - Centrum Alergologii Teresa Hofman Sp. Z o.o., Poznan
  - RCMed Oddz. Sochaczew, Sochaczew
  - Centrum Medyczne Lucyna Andrzej Dymek, Strzelce Opolskie
  - Alergo-Med Specjalistyczna Przychodnia Lekarska, Tarnów
- Ukraine (17):
  - Chernihiv City Hospital #2, Therapy Department, Chernihiv
  - Medical and Sanitary Unit of Private Joint Stock Company Kharkiv Tractor Plant, Therapeutic Department, Kharkiv Medical Academy of Postgraduate Education, Chair of General Practice-family Medicine, Kharkiv
  - Communal Non-Commercial Enterprize of Kharkiv Regional Council Regional Clinical Hospital, Pulmonary-Allergological Department with Immunological and Therapeutic Beds, Kharkiv
  - City Clinical Hospital #13, Kharkiv
  - Communal Non-profit Enterprise "Kherson City Clinical Hospital named after Ye. Ye. Karabelesh" of the Kherson City Council, Pulmonary Therapeutic Department, Kherson
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv
  - Medical Center of Edelweiss Medics LLC , Treatment and Prevention Department, Kyiv
  - Municipal Non-commercial Enterprise "Consultative-Diagnostics Center" of Desnyanskyi District of Kyiv, Therapy Department, Kyiv
  - Medical Center of LLC Medbud-Clinic, Treatment and Prevention Department, Kyiv
  - National Institute of Phthisiology and Pulmonology, Department of Pulmonology, Kyiv
  - SI "National Institute of Phthisiology and Pulmonology n.a. F.G.Yanovskyi under NAMS of Ukraine," Department of Diagnostic, Therapy and Clinical Pharmacology of Lung Diseases, Kyiv
  - Kyiv Railway Clinical Hospital No2 of Branch Health Center of the JSC Ukrainian Rail, Department of Pulmonology, Kyiv
  - Clinic of SI National Research Centre of Radiation Medicine of NAMS of Ukraine, Unit of Pulmonology of Department of Therapy of Radiation Consequences of Clinical Radiology Institute, Kyiv
  - Municipal Enterprise Volyn Regional Clinical Hospital of Volyn Regional Council, Pulmonology Department, Lutsk
  - The 1st City Clinical Hospital of Poltava City Council, Poltava
  - Small Business Private Enterprise Medical Centre "Pulse", Therapeutic Department, Vinnytsia
  - CNE Vinnytsia Regional Clinical Hospital named after N.I. Pirogov VRC, Regional Treatment and Diagnostic Pulmonology Center, Chair of Internal Medicine #1, Vinnytsia National Medical University n.a.M.I.Pyrogov, Vinnytsia
- United Kingdom (11):
  - Respiratory Clinical Trials, Cottingham, East Yorkshire
  - Wythenshawe Hospital, Manchester, Greater Manchester
  - MeDiNova South London Quality Research Site, Sidcup, Kent
  - BMI Bishops Wood Hospital, Northwood, Middlesex
  - MeDiNova North London Quality Research Site, Northwood, Middlesex
  - Medinova Research Northamptonshire Quality Research Site, Corby, Northamptonshire
  - Northumbria Healthcare NHS Foundation Trust, North Tyneside General Hospital, North Shields, Northumberland
  - Medinova Yorkshire Quality Research Site, Bradford, West Yorkshire
  - Belfast City Hospital, Belfast
  - Kings College Hospital, London
  - West Walk Surgery, Yate

REFERENCES:
- [Derived] McGarvey L, Smith JA, Morice A, Birring SS, Chung KF, Dicpinigaitis PV, Niimi A, Benninger MS, Sher M, Matsunaga Y, Miyazaki S, Machida M, Ishihara H, Mahmood A, Gomez JC. A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase 2b Trial of P2X3 Receptor Antagonist Sivopixant for Refractory or Unexplained Chronic Cough. Lung. 2023 Feb;201(1):25-35. doi: 10.1007/s00408-022-00592-5. Epub 2022 Dec 13. PMID 36512069

RESULTS

PARTICIPANT FLOW:
Groups:
- S-600918 50 mg: Participants received 50 mg S-600918 tablets orally once daily for 28 days
- S-600918 150 mg: Participants received 150 mg S-600918 tablets orally once daily for 28 days
- S-600918 300 mg: Participants received 300 mg S-600918 tablets orally once daily for 28 days
- Placebo: Participants received placebo tablets orally once daily for 28 days
Period: Overall Study
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Started | 101 | 103 | 100 | 102
Received At Least 1 Dose of Study Drug | 100 | 103 | 100 | 102
Completed | 100 | 99 | 92 | 99
Not Completed | 1 | 4 | 8 | 3
Not completed — COVID-19 reason other than AE | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 0
Not completed — Adverse Event | 1 | 1 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug and who had cough monitor assessment at both baseline and at least 1 visit after initiation of study drug administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo | Total
Number analyzed (Participants) | 100 | 102 | 96 | 102 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11.2) | 57.2 (12.5) | 56.1 (12.4) | 56.1 (11.5) | 57.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 65 | 77 | 295
  Male | 22 | 27 | 31 | 25 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 4 | 2 | 14
  Not Hispanic or Latino | 95 | 98 | 92 | 100 | 385
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Asian | 25 | 25 | 25 | 22 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 4 | 9
  White | 71 | 76 | 69 | 72 | 288
  More than one race | 1 | 0 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Average Coughs per Hour in 24 Hours [Mean (Standard Deviation); unit: number of coughs] | 30.40 (22.92) | 40.95 (64.68) | 36.21 (37.91) | 33.85 (34.60) | 35.36 (43.00)
Weekly Severity of Cough [Mean (Standard Deviation); unit: score on a scale] — Baseline cough severity was assessed by the participant by a visual analog scale, with scores ranging from 0 to 100. Higher scores indicated higher cough severity.
  score on a scale | 74.8 (14.0) | 73.6 (13.8) | 72.6 (15.3) | 71.6 (14.5) | 73.1 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Number of Coughs Per Hour in 24 Hours Following 4 Weeks of Study Treatment
Description: Change in cough was calculated based upon the number of coughs per hour in 24 hours at Week 4 and baseline. Results are presented as percent change from baseline. Reported percent change is based on a mixed model for the log-transformed ratio of the number of coughs per hour in 24 hours at each visit with treatment, week, and treatment-by-week as fixed effect, participant as random effect, and region (Japan, Europe, or the United States) and the log-transformed coughs per hour in 24 hours at baseline as covariates. The number of coughs per hour while awake was measured using a cough monitor.
Time Frame: Baseline to Week 4
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug and who had cough monitor assessment at both baseline and at least 1 visit after initiation of study drug administration. Here 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 87 | 95
percentage change | -55.16 [-62.80 to -45.94] | -61.08 [-67.71 to -53.08] | -65.32 [-71.37 to -57.99] | -60.38 [-67.07 to -52.32]
Statistical Analysis 1: Comparison: S-600918 50 mg vs S-600918 150 mg vs S-600918 300 mg vs Placebo; The null hypotheses of equality between the treatment and placebo effects were tested using a mixed model, containing treatment group, week, and interaction between treatment groups and week as fixed effects; participant as random effect; and region and the common logarithm of the frequency of coughs per hour at baseline as covariates. Covariance structure was given as unstructured; Test type: Equivalence — Placebo (N = 102) vs S-600918 50 mg, 150 mg, 300 mg; p = 0.9334, ANCOVA — P-value was evaluated at the 2-sided alpha level of 0.05

2. Secondary Outcome: Number of Participants With 30%, 50%, and 70% Reduction in Number of Coughs Per Hour Over 24 Hours After 4 Weeks of Study Treatment
Description: The number of coughs per hour for 24 hours was measured using a cough monitor.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 87 | 95
Participants
  ≥ 30% Reduction | 55 | 66 | 66 | 61
  ≥ 50% Reduction | 38 | 46 | 50 | 49
  ≥ 70% Reduction | 24 | 26 | 31 | 27

3. Secondary Outcome: Percent Change in Number of Coughs Per Hour While Awake Following 4 Weeks of Study Treatment
Description: Change in cough was calculated based upon the number of coughs per hour in 24 hours at Week 4 and baseline. Results are presented as percent change from baseline. Reported percent change is based on a mixed model for the log-transformed ratio of the number of coughs per hour while awake at each visit with treatment, week, and treatment-by-week as fixed effect, participants as random effect, and region and the log-transformed coughs per hour while awake at baseline as covariates. The number of coughs per hour while awake was measured using a cough monitor.
Time Frame: Baseline to Week 4
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug and who had cough monitor assessment at both baseline and at least 1 visit after initiation of study drug administration. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure at the specified timeframe.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage change
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 87 | 95
percentage change | -55.77 [-63.61 to -46.25] | -61.75 [-68.52 to -53.52] | -66.33 [-72.43 to -58.89] | -60.31 [-62.27 to -51.87]

4. Secondary Outcome: Number of Participants With 30%, 50% and 70% Reduction in Number of Coughs Per Hour While Awake After 4 Weeks of Study Treatment
Description: The number of coughs per hour while awake was measured using a cough monitor.
Time Frame: Baseline to Week 4
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug and who had cough monitor assessment at both baseline and at least 1 visit after initiation of study drug administration. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants evaluable at the specified timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 92 | 89 | 87 | 95
Participants
  ≥ 30% Reduction | 55 | 67 | 67 | 61
  ≥ 50% Reduction | 41 | 48 | 51 | 46
  ≥ 70% Reduction | 22 | 26 | 29 | 25

5. Secondary Outcome: Percent Change in Number of Coughs Per Hour While Asleep Following 4 Weeks of Study Treatment
Description: Change in cough was calculated based upon the number of coughs per hour in 24 hours at Week 4 and baseline. Results are presented as percent change from baseline. Reported percent change is based on a mixed model for the log-transformed ratio of the number of coughs per hour while asleep at each visit with treatment, week, and treatment-by-week as fixed effect, participants as random effect, and region and the log-transformed coughs per hour while asleep at baseline as covariates. The number of coughs per hour while awake was measured using a cough monitor.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percentage change
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 92 | 87 | 86 | 93
percentage change | -54.43 [-66.61 to -37.80] | -53.17 [-65.89 to -35.73] | -65.48 [-74.96 to -52.41] | -52.73 [-65.30 to -35.61]

6. Secondary Outcome: Change From Baseline in Weekly Cough Severity Following 4 Weeks of Study Treatment
Description: Cough severity was assessed by the participant by a visual analog scale with numbers from 0 to 100. Results are presented as change from baseline. Reported change is based on a mixed model for the change in weekly cough severity score after 4 weeks of treatment with treatment, week, and treatment-by-week as fixed effect, participant as random effect, and region (Japan, Europe, or the United States) and the severity score at baseline as covariates. Higher scores indicated higher cough severity.
Time Frame: Baseline to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 93 | 92 | 91 | 93
score on a scale | -19.99 [-24.47 to -15.51] | -22.95 [-27.42 to -18.47] | -28.29 [-32.86 to -23.72] | -21.74 [-26.20 to -17.27]

7. Secondary Outcome: Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score
Description: The LCQ is a patient-reported quality of life (QOL) measure of chronic cough. The questionnaire consists of 19 items to which the participant responds on a 7-point Likert response scale (from 1 to 7). Each item assesses symptoms during cough and the effect of cough on 3 main domains: physical, psychological and social. Domain scores range from 1-7, and the total score ranges from 3 - 21. Higher score indicates a better quality of life. Results are presented as change from baseline. Reported change is based on a mixed model for the change in LCQ Total Score after 4 weeks of treatment with treatment, week, and treatment-by-week as fixed effect, participant as random effect, and region (Japan, Europe, or the United States) and the LCQ Score of corresponding domain at baseline as covariates.
Time Frame: Baseline to Week 4
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 86 | 82 | 78 | 82
score on a scale | 2.80 [2.17 to 3.43] | 3.10 [2.46 to 3.75] | 3.86 [3.19 to 4.53] | 3.17 [2.52 to 3.82]

8. Secondary Outcome: Number of Responders Defined as Participants With an Increase in LCQ of ≥ 1.3 Points
Description: The LCQ is a patient-reported quality of life (QOL) measure of chronic cough. The questionnaire consists of 19 items to which the participant responds on a 7-point Likert response scale (from 1 to 7). Each item assesses symptoms during cough and the effect of cough on 3 main domains: physical, psychological and social. Domain scores range from 1-7, and the total score ranges from 3 - 2. A higher score indicates a better quality of life.
Time Frame: Baseline to Week 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 86 | 82 | 78 | 82
Participants | 53 | 56 | 60 | 48

9. Secondary Outcome: Change From Baseline in International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF)
Description: The ICIQ-SF is a questionnaire used to evaluate the frequency, severity, and impact of urinary incontinence on the quality of life. The questionnaire includes 3 items with responses measured on Likert scales, and 1 item that is measured via a qualitative response. The 3 nominal responses are summed to give the ICIQ score (this total ICIQ-SF score can range from 0 to 21), where a higher score indicates more severe symptoms. The 1 item remaining that is measured via qualitative response is not given a score; rather, the participant selects 1 description out of 8 possible descriptions of this item.
Time Frame: Baseline to Week 4
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug and who had cough monitor assessment at both baseline and at least 1 visit after initiation of study drug administration. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure and 'Number analyzed' = participants evaluable at the specified timeframe for this specific outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 99 | 101 | 96 | 102
score on a scale
  Baseline, Female With Symptoms: number analyzed (Participants) | 52 | 47 | 41 | 53
  Baseline, Female With Symptoms | 9.9 (5.0) | 8.8 (5.2) | 9.2 (4.6) | 8.6 (4.2)
  Change at Week 4 - Female With Symptoms: number analyzed (Participants) | 49 | 42 | 38 | 49
  Change at Week 4 - Female With Symptoms | -2.2 (3.9) | -1.2 (3.4) | -1.6 (3.8) | -1.2 (3.3)
  Baseline, Female Without Symptoms: number analyzed (Participants) | 25 | 27 | 24 | 24
  Baseline, Female Without Symptoms | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Change at Week 4 - Female Without Symptoms: number analyzed (Participants) | 23 | 24 | 23 | 20
  Change at Week 4 - Female Without Symptoms | 0.9 (2.2) | 0.1 (0.4) | 0.5 (1.3) | 0.3 (1.1)
  Baseline, Male With Symptoms: number analyzed (Participants) | 4 | 7 | 6 | 7
  Baseline, Male With Symptoms | 9.5 (5.3) | 5.0 (2.3) | 6.7 (4.0) | 5.0 (2.2)
  Change at Week 4 - Male With Symptoms: number analyzed (Participants) | 4 | 7 | 5 | 7
  Change at Week 4 - Male With Symptoms | -2.0 (8.3) | -0.7 (2.7) | -1.0 (2.3) | -0.9 (2.2)
  Baseline, Male Without Symptoms: number analyzed (Participants) | 18 | 20 | 25 | 18
  Baseline, Male Without Symptoms | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Change at Week 4 - Male Without Symptoms: number analyzed (Participants) | 16 | 19 | 25 | 15
  Change at Week 4 - Male Without Symptoms | 0.8 (2.4) | 1.3 (3.2) | 0.5 (1.4) | 0.0 (0.0)

10. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36)
Description: The SF-36 is a 36-item questionnaire to assesses a participant's health status using 8 health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. The mental component reports the average of all the emotionally relevant items and the physical component reports the average of all the physically relevant items. Each component is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 indicates no disability. Median change can range from -100 to 100. A positive median change indicates an improved outcome.
Time Frame: Baseline to Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 99 | 101 | 96 | 102
score on a scale
  Baseline - Physical Component Score | 38.4 (6.3) | 38.6 (5.7) | 38.1 (5.6) | 37.8 (5.5)
  Change at Week 4 - Physical Component Score: number analyzed (Participants) | 92 | 91 | 91 | 91
  Change at Week 4 - Physical Component Score | -0.3 (5.0) | -0.9 (4.5) | -0.9 (4.6) | -1.3 (5.0)
  Baseline - Mental Component Score | 46.1 (10.3) | 47.1 (9.0) | 47.5 (8.7) | 47.2 (9.2)
  Change at Week 4 - Mental Component Score: number analyzed (Participants) | 92 | 91 | 91 | 91
  Change at Week 4 - Mental Component Score | 2.2 (5.9) | 1.9 (6.0) | 2.6 (6.0) | 3.3 (6.0)

11. Secondary Outcome: Number of Responders as Assessed by Patient Global Impression of Change (PGIC)
Description: The PGIC is a patient-reported measure of overall health status and consists of 1 item adapted from the Clinical Global Impressions scale. The participant selects 1 description out of 7 possible descriptions of this item. The descriptions are numbered from 1 through 7, where lower numbers indicate better quality of life. Participants were considered responders if they reported "Very much improved", "Much improved", or "Minimally improved" from baseline on the PGIC assessment.
Time Frame: Week 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
Number analyzed (Participants) | 100 | 102 | 96 | 102
Participants | 57 | 72 | 79 | 65

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | S-600918 50 mg | S-600918 150 mg | S-600918 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/103 | 0/100 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/103 | 0/100 | 0/102
Other Adverse Events (participants affected / at risk) | 5/101 | 15/103 | 34/100 | 10/102
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | S-600918 50 mg (N=101) | S-600918 150 mg (N=103) | S-600918 300 mg (N=100) | Placebo (N=102)
Dysgeusia (Nervous system disorders) | 2 | 12 | 27 | 3
Headache (Nervous system disorders) | 3 | 2 | 1 | 7
Hypogeusia (Nervous system disorders) | 0 | 1 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04110054/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04110054/SAP_001.pdf